CLINICAL TRIAL: NCT02093663
Title: A Phase 3, Multicenter, Randomized, Double-blind Study to Determine the Safety and Efficacy of MMX Mesalamine/Mesalazine in Pediatric Subjects With Mild to Moderate Ulcerative Colitis, in Both Acute and Maintenance Phases
Brief Title: Safety and Efficacy of MMX Mesalamine/Mesalazine in Pediatric Subjects With Mild to Moderate Ulcerative Colitis
Acronym: PACE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD476-319; 2013-001744-65 (EudraCT Number)
Record Dates: First submitted 2014-03-17; First posted 2014-03-21 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Ulcerative Colitis
Keywords: Mild; Moderate
MeSH Terms: conditions — Colitis, Ulcerative; Lymphoma, Follicular | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- MMX Mesalamine/Mesalazine (Low Dose) (Experimental): Once daily, tablets - the amount depends on the participants weight; 900 milligram per day (mg/day) for participants weighing 18 kg to less than or equal to (<=) 23 kilograms (kg); 1200 mg/day for participants weighing greater than (>) 23 kg to <= 35 kg; 1800 mg/day for participants weighing > 35 kg to <= 50 kg; 2400 mg/day for participants weighing > 50 kg to <= 90 kg.
  Interventions: Drug: MMX Mesalamine/Mesalazine (Low Dose)
- MMX Mesalamine/Mesalazine (High Dose) (Experimental): Once daily, tablets - the amount depends on the participants weight;1800 mg/day for participants weighing 18 kg to <= 23 kg; 2400 mg/day for participants weighing > 23 kg to <= 35 kg; 3600 mg/day for participants weighing > 35 kg to <= 50 kg; 4800 mg/day for participants weighing > 50 kg to <= 90 kg.
  Interventions: Drug: MMX Mesalamine/Mesalazine (High Dose)

INTERVENTIONS:
Drug: MMX Mesalamine/Mesalazine (Low Dose) — Once daily, tablets - the amount depends on the participants weight; 900 milligram per day (mg/day) for participants weighing 18 kg to less than or equal to (<=) 23 kilograms (kg); 1200 mg/day for participants weighing greater than (>) 23 kg to <= 35 kg; 1800 mg/day for participants weighing > 35 kg to <= 50 kg; 2400 mg/day for participants weighing > 50 kg to <= 90 kg.
  Other Names: Lialda; Mezavant
  Arms: MMX Mesalamine/Mesalazine (Low Dose)
Drug: MMX Mesalamine/Mesalazine (High Dose) — Once daily, tablets - the amount depends on the participants weight;1800 mg/day for participants weighing 18 kg to <= 23 kg; 2400 mg/day for participants weighing > 23 kg to <= 35 kg; 3600 mg/day for participants weighing > 35 kg to <= 50 kg; 4800 mg/day for participants weighing > 50 kg to <= 90 kg.
  Other Names: Mezavant; Lialda
  Arms: MMX Mesalamine/Mesalazine (High Dose)

SUMMARY:
To assess clinical response to MMX mesalamine/mesalazine between a low and high dose in children and adolescents aged 5-17 years with mild to moderate Ulcerative Colitis (UC) or who are in remission.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to voluntarily provide written, signed, and dated (personally or via a legally authorized representative [LAR]) informed consent or assent as applicable to participate in the study.
2. Subject's parent/LAR demonstrates an understanding, ability, and willingness to fully comply with study procedures and restrictions.
3. Male and female children and adolescents aged 5-17 years, inclusive.
4. Body weight 18-90kg.
5. Male, or non-pregnant, non-lactating female who agrees to comply with any applicable contraceptive requirements of the protocol or females of non-childbearing potential.
6. Diagnosed with mild to moderate UC, established by sigmoidoscopy or colonoscopy with compatible histology. Screened subjects may also have an unconfirmed diagnosis of mild to moderate UC; however the diagnosis of mild to moderate UC must have been established by sigmoidoscopy or colonoscopy with compatible histology prior to baseline visit.
7. Subject is able to swallow the investigational product whole.

   Double-blind Acute Phase:
8. Partial UC-DAI score ≥2 (a combined rectal bleeding and stool frequency score ≥1 and PGA=1 or 2) at the Baseline Visit, for which 5-ASA would be used as part of normal treatment.
9. If the subject is on 5-ASA treatment prior to study entry, then the dose must be stable. Stable therapy is defined as no change in dose, or no initiation of 5-ASA, from the onset of the current acute flare through discontinuation of therapy (required at the Baseline Visit).

   Double-blind Maintenance Phase:
10. Partial UC-DAI ≤1 (rectal bleeding=0, stool frequency ≤1, and PGA=0) at the Baseline Visit.

Exclusion Criteria:

1. Severe UC (defined by PGA=3).
2. Crohn's disease, bleeding disorders, active peptic ulcer disease, or UC known to be confined to the rectum (isolated rectal proctitis).
3. Asthma, only if known to be 5 ASA sensitive.
4. Positive stool culture for enteric pathogens (including Salmonella, Shigella, Yersinia, Aeromonas, Plesiomonas, or Campylobacter). Clostridium difficile toxin, ova, or parasites present.
5. Systemic or rectal corticosteroid use within 4 weeks prior to the Screening Visit. Topical, intranasal, or inhaled use is not exclusionary.
6. Immunomodulator (6-mercaptopurine, azathioprine) use within 6 weeks prior to the Screening Visit.
7. History of biologic (eg, anti-tumor necrosis factor agents, integrin receptor antagonists) use at any time.
8. Antibiotic use within 7 days prior to the Screening Visit.
9. Any anti-inflammatory drugs, not including 5-ASA treatment but including non-steroidal anti-inflammatory drugs such as aspirin, COX-2 inhibitors or ibuprofen, within 7 days prior to the Screening Visit unless used at over-the-counter levels for <3 days. However, prophylactic use of a stable dose of aspirin up to 325mg/day for cardiac disease is permitted.
10. Prebiotic/probiotic use within 7 days prior to the Screening Visit. Yogurt products are permitted.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 107 (Actual)
Dates: Start 2014-12-12 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shire Director, Study Director — Takeda
Locations (33):
- United States (9):
  - University of Maryland Children's Hospital, Baltimore, Maryland
  - John Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Newton Wellesley Hospital, Newton, Massachusetts
  - University of Minnesota Children's Hospital, Minneapolis, Minnesota
  - Mayo Clinic Gastroenterology, Rochester, Minnesota
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Carilion Medical Center, Roanoke, Virginia
- University of Alberta Pediatric Gastroenterology & Nutrition, Edmonton, Alberta, Canada
- Hungary (5):
  - Szent Janos Korhaz És Észak-budai Egyesitett Korha, Budapest
  - Bekes Megyei Pandy Kalman Korhaz, Gyula
  - Baz Megyei Korhaz Es Egyetemi Oktatokorhaz, Miskolc
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktato Korhaz, Nyíregyháza
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- Israel (4):
  - Soroka Medical Center, Beersheba
  - Rambam Health Corporation, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Schneider Medical Centre, Petah Tikva
- Poland (7):
  - Uniwersytecki Dzieciecy Szpital Kliniczny im. Ludwika Zamenhofa, Bialystok
  - Klinika Pediatrii Gastroenterologii I Zywienia, Krakow
  - Klinika Gastroenterologii I Pediatrii, Lodz
  - Wojewodzki Specjalistyczny Szpital Dzieciecy, Olsztyn
  - Gabinet Lekarski-Bartosz Korczowski, Rzeszów
  - Oddzial Gastroenterologii I Hepatologii, Warsaw
  - Uniwersytecki Szpital Kliniczny We Wrocławiu, Wroclaw
- Slovakia (3):
  - Detská fakultná nemocnica s poliklinikou, Banská Bystrica
  - University Children's Hospital, Bratislava
  - Univerzitna Nemocnica Martin, Martin
- United Kingdom (4):
  - Alder Hey Children's Hospital, Liverpool
  - Barts Health NHS Trust, Royal London Hospital, London
  - King's College Hospital, London
  - Great Ormond Street Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Croft NM, Korczowski B, Kierkus J, Caballero B, Thakur MK. Safety and efficacy of multimatrix mesalamine in paediatric patients with mild-to-moderate ulcerative colitis: a phase 3, randomised, double-blind study. EClinicalMedicine. 2023 Oct 6;65:102232. doi: 10.1016/j.eclinm.2023.102232. eCollection 2023 Nov. PMID 37855022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 50 study centers and 33 sites consented at least 1 participant between 12 December 2014 (first participant first visit) and 28 November 2018 (last participant last visit).
Pre-assignment Details: Study was conducted in three phases as double blind acute (DBA), open label acute (OLA), and double blind maintenance (DBM) phase. Overall, 107 participants were enrolled and entered into DBA or DBM directly and eligible participants entered into DBM phase after DBA or OLA through DBA. Total, 105 participants received treatment and 65 completed.
Groups:
- Double-Blind Acute (DBA) Phase: Low Dose: Participants with partial UC-DAI > or =2 and mucosal appearance = 2 or 3 entered the DBA phase. During the DBA low dose phase participants weighing 18 to < or =23 kg, >23 to < or =35 kg, > 35 to < or =50 kg, > 50 to < or =90 kg received 900, 1200, 1800, and 2400 mg/day of MMX mesalamine/mesalazine tablet orally once daily for 8 weeks respectively.
- Double-Blind Acute (DBA) Phase: High Dose: Participants with partial UC-DAI > or =2 and mucosal appearance = 2 or 3 entered the DBA phase. During the DBA high dose phase participants weighing 18 to < or =23 kg, > 23 to < or =35 kg, > 35 to < or =50 kg, > 50 to < or =90 kg received 1800, 2400, 3600, and 4800 mg/day of MMX mesalamine/mesalazine tablet orally once daily for 8 weeks respectively.
- Open-Label Acute Phase (OLA): High Dose: During the OLA High dose phase participants weighing 18 to <=23 kg, > 23 to < or =35 kg, >35 to < or = 50 kg, > 50 to < or = 90 kg received 1800, 2400, 3600, and 4800 mg/day of MMX mesalamine/mesalazine tablet orally once daily for 8 weeks respectively.
- Double-Blind Maintenance (DBM) Phase: Low Dose: Participants with partial UC-DAI < or =1 and mucosal appearance = 0 or 1 entered the DBM phase directly. Also, participants with a clinical response (partial UC-DAI < or =1) after completion of DBA phase or OLA phase entered into the DBM phase. During the DBM low dose phase participants weighing 18 to < or =23 kg, > 23 to < or =35 kg, > 35 to < or =50 kg, > 50 to < or =90 kg received 900, 1200, 1800, and 2400 mg/day of MMX mesalamine/mesalazine tablet orally once daily for 26 weeks respectively.
- Double-Blind Maintenance (DBM) Phase: High Dose: Participants with partial UC-DAI < or =1 and mucosal appearance = 0 or 1 entered the DBM phase directly. Also, participants with a clinical response (partial UC-DAI < or =1) after completion of DBA phase or OLA phase entered into the DBM phase. During the DBM high dose phase participants weighing 18 to <=23 kg, > 23 to < or =35 kg, >35 to < or = 50 kg, > 50 to < or = 90 kg received 1800, 2400, 3600, and 4800 mg/day of MMX mesalamine/mesalazine tablet orally once daily for 26 weeks respectively.
Period: Double Blind Acute Phase (8 Weeks)
Arm/Group | Double-Blind Acute (DBA) Phase: Low Dose | Double-Blind Acute (DBA) Phase: High Dose | Open-Label Acute Phase (OLA): High Dose | Double-Blind Maintenance (DBM) Phase: Low Dose | Double-Blind Maintenance (DBM) Phase: High Dose
Started | 27 | 26 | 0 | 0 | 0
Completed | 19 | 22 | 0 | 0 | 0
Not Completed | 8 | 4 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 5 | 0 | 0 | 0 | 0
Not completed — Subjects who Continued in the Study | 2 | 4 | 0 | 0 | 0
Period: Open Label Acute Phase (8 Weeks)
Arm/Group | Double-Blind Acute (DBA) Phase: Low Dose | Double-Blind Acute (DBA) Phase: High Dose | Open-Label Acute Phase (OLA): High Dose | Double-Blind Maintenance (DBM) Phase: Low Dose | Double-Blind Maintenance (DBM) Phase: High Dose
Started | 0 | 0 | 18 | 0 | 0
Participants Entered OLA Via DBA | 0 | 0 | 18 | 0 | 0
Completed | 0 | 0 | 12 | 0 | 0
Not Completed | 0 | 0 | 6 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 5 | 0 | 0
Period: Double Blind Maintenance Phase(26 Weeks)
Arm/Group | Double-Blind Acute (DBA) Phase: Low Dose | Double-Blind Acute (DBA) Phase: High Dose | Open-Label Acute Phase (OLA): High Dose | Double-Blind Maintenance (DBM) Phase: Low Dose | Double-Blind Maintenance (DBM) Phase: High Dose
Started | 0 | 0 | 0 | 42 | 45
Participants Entered Directly to DBM | 0 | 0 | 0 | 26 | 26
Participants Entered DBM Via DBA | 0 | 0 | 0 | 12 | 15
Participants Entered DBM Via OLA | 0 | 0 | 0 | 4 | 4
Completed | 0 | 0 | 0 | 32 | 34
Not Completed | 0 | 0 | 0 | 10 | 11
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 6 | 7
Not completed — Other (unspecified) | 0 | 0 | 0 | 1 | 1
Not completed — Missing | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisted of randomized participants who had taken at least 1 dose of investigational product. Few participants had multiple movement within the arms of the study at different levels and unique participants baseline was not analysed, only overall participant data was planned, analysed and reported to avoid double-counting.
Groups:
- Overall Study: Participants with partial UC-DAI > or =2 and mucosal appearance = 2 or 3 entered the DBA phase; with UC-DAI between 1 and 2 entered the OLA phase, after completing DBA phase; with UC-DAI < or = 1 and mucosal appearance = 0 or 1 entered the DBM phase directly. Also, participants who had a clinical response (partial UC-DAI < or =1) after completion of DBA phase or OLA phase entered into the DBM phase. During the DBA and DBM phase, participants received 900 to 2400 mg/day (low dose) and 1800 to 4800 mg/day (high dose) of MMX mesalamine/mesalazine tablet orally once daily for 8 and 26 weeks respectively. During OLA phase, participants received the high dose for 8 weeks.
Arm/Group | Overall Study
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (2.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 104
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 101
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response During Double-Blind Acute Phase at Week 8
Description: Clinical response was defined as partial ulcerative colitis disease activity index (UC-DAI) score < or =1 with rectal bleeding = 0, stool frequency < or =1, and physician's global assessment (PGA = 0). Number of participants with clinical response were reported.
Time Frame: Week 8
Population: Double-blind acute phase safety analysis set consisted of randomized participants who had taken at least 1 dose of investigational product during the double-blind acute phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Acute (DBA) Phase: Low Dose | Double-Blind Acute (DBA) Phase: High Dose
Number analyzed (Participants) | 27 | 26
Participants | 10 | 17
Statistical Analysis 1: Comparison: Double-Blind Acute (DBA) Phase: Low Dose vs Double-Blind Acute (DBA) Phase: High Dose; This study is not powered to detect differences between treatment groups and other sensitivity analysis (last observation carried forward [LOCF] and complete case) intended to examine the robustness of the treatment estimate. This was an estimation study, and p-values were presented as descriptive statistics; Test type: Other; p = 0.039, Uncorrected Chi-squared Test; Odds Ratio (OR) = 3.21, 95% CI 2-sided [1.04 to 9.88]

2. Primary Outcome: Number of Participants With Clinical Response During Double-blind Maintenance Phase at Week 26
Description: Clinical response was defined as partial UC-DAI <=1 with (rectal bleeding = 0, stool frequency < or =1, and PGA = 0). Number of participants who had maintained clinical response were reported.
Time Frame: Week 26
Population: Double-blind maintenance phase safety analysis set consisted of randomized participants who had taken at least 1 dose of investigational product during the double-blind maintenance phase.
Measure: Count of Participants; unit: Participants
Groups:
- Double-Blind Maintenance (DBM) Phase: Low Dose: Participants with partial UC-DAI < or =1 and mucosal appearance = 0 or 1 entered the DBM phase directly. Also, participants with a clinical response (partial UC-DAI < or =1) after completion of DBA phase or OLA phase entered into the DBM phase. During the DBM low dose phase participants weighing 18 to <=23 kg, >23 to <=35 kg, >35 to < or =50 kg, >50 to < or =90 kg received 900, 1200, 1800, and 2400 mg/day of MMX mesalamine/mesalazine tablet orally once daily for 26 weeks respectively.
- Double-Blind Maintenance (DBM) Phase: High Dose: Participants with partial UC-DAI < or =1 and mucosal appearance = 0 or 1 entered the DBM phase directly. Also, participants with a clinical response (partial UC-DAI < or =1) after completion of DBA phase or OLA phase entered into the DBM phase. During the DBM high dose phase participants weighing 18 to <=23 kg, >23 to <=35 kg, >35 to < or =50 kg, >50 to < or =90 kg received 1800, 2400, 3600, and 4800 mg/day of MMX mesalamine/mesalazine tablet orally once daily for 26 weeks respectively.
Arm/Group | Double-Blind Maintenance (DBM) Phase: Low Dose | Double-Blind Maintenance (DBM) Phase: High Dose
Number analyzed (Participants) | 42 | 45
Participants | 23 | 24
Statistical Analysis 1: Comparison: Double-Blind Maintenance (DBM) Phase: Low Dose vs Double-Blind Maintenance (DBM) Phase: High Dose; This study is not powered to detect differences between treatment groups and other sensitivity analysis (LOCF and complete case) intended to examine the robustness of the treatment estimate. This was an estimation study, and p-value s were presented as descriptive statistics; Test type: Other; p = 0.981, Cochran-Mantel-Haenszel — P-value were based on a Cochran-Mantel-Haenszel test stratified by prior response status; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.42 to 2.34]

3. Secondary Outcome: Number of Participants With Clinical and Endoscopic Response During Double Blind Acute Phase at Week 8 Using Central Reading
Description: Clinical and endoscopic response was defined as UC-DAI <=2 with rectal bleeding = 0 and stool frequency <=1, and PGA = 0, and with mucosal healing (endoscopy score <=1) at least a 1 point reduction in endoscopy score from baseline based on central reading. Participants with missing data at week 8 were assumed not to had a clinical response. Participants who completed week 8 but did not have central reading endoscopies at both baseline and week 8 were excluded. Number of participants with clinical and endoscopic response were reported.
Time Frame: Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Double-Blind Acute (DBA) Phase: Low Dose: Participants with partial UC-DAI > or =2 and mucosal appearance = 2 or 3 entered the DBA phase. During the DBA low dose phase participants weighing 18 to < or =23 kg, > 23 to < or =35 kg, > 35 to < or =50 kg, > 50 to < or =90 kg received 900, 1200, 1800, and 2400 mg/day of MMX mesalamine/mesalazine tablet orally once daily for 8 weeks respectively.
Arm/Group | Double-Blind Acute (DBA) Phase: Low Dose | Double-Blind Acute (DBA) Phase: High Dose
Number analyzed (Participants) | 27 | 26
Participants | 1 | 3
Statistical Analysis 1: Comparison: Double-Blind Acute (DBA) Phase: Low Dose vs Double-Blind Acute (DBA) Phase: High Dose; This study is not powered to detect differences between treatment groups and other sensitivity analysis (LOCF and complete case) intended to examine the robustness of the treatment estimate. This was an estimation study, and p-values were presented as descriptive statistics; Test type: Other; p = 0.400, Fisher Exact — P-value was calculated based on Fisher's exact test; Difference in proportions = 50.0, 95% CI 2-sided [-19.3 to 100.0]

4. Secondary Outcome: Number of Participants With Clinical and Endoscopic Response During Double Blind Acute Phase at Week 8 Using Local Reading
Description: Clinical and endoscopic response was defined as UC-DAI < or =2 with rectal bleeding = 0 and stool frequency < or =1, and PGA = 0, and with mucosal healing (endoscopy score < or =1) at least a 1 point reduction in endoscopy score from baseline based on local reading. Participants with missing data at week 8 were assumed not to had a clinical response. Participants who completed week 8 but did not have local reading endoscopies at both baseline and week 8 were excluded. Number of participants with clinical and endoscopic response were reported.
Time Frame: Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Acute (DBA) Phase: Low Dose | Double-Blind Acute (DBA) Phase: High Dose
Number analyzed (Participants) | 27 | 26
Participants | 1 | 4
Statistical Analysis 1: Comparison: Double-Blind Acute (DBA) Phase: Low Dose vs Double-Blind Acute (DBA) Phase: High Dose; This study is not powered to detect differences between treatment groups and other sensitivity analysis (LOCF and complete case) intended to examine the robustness of the treatment estimate; Test type: Other; p = 0.333, Fisher Exact — P-value was based on a Fisher's exact test; Difference in proportions = 50.0, 95% CI 2-sided [-19.3 to 100.0]

5. Secondary Outcome: Change From Baseline in Daily Ulcerative Colitis Scale (DUCS) Score During Double-Blind Acute Phase
Description: DUCS score was to measure 7 specific signs or symptom and one impact (abdominal pain, nocturnal stool, daytime stool, blood in stool, diarrhea, urgency, tiredness) of UC with each item score ranged from 0 (worst) to 10 (best) with the overall score ranged from 0 (worst) to 70 (best) based on the responses. Change in the DUCS score from baseline to Week 8 during DBA phase were reported.
Time Frame: Baseline to Week 8
Population: Double-blind acute phase safety analysis set consisted of randomized participants who had taken at least 1 dose of investigational product during the double-blind acute phase. Here, number of participants analyzed signifies participants who were evaluable for this measure category.
Measure: Mean (Standard Error); unit: Score on the scale
Arm/Group | Double-Blind Acute (DBA) Phase: Low Dose | Double-Blind Acute (DBA) Phase: High Dose
Number analyzed (Participants) | 27 | 26
Score on the scale
  Baseline | 32.2 (2.86) | 31.6 (2.88)
  Week 2: number analyzed (Participants) | 24 | 23
  Week 2 | -14.1 (3.80) | -13.2 (3.50)
  Week 4: number analyzed (Participants) | 20 | 22
  Week 4 | -15.6 (3.96) | -16.7 (4.01)
  Week 8: number analyzed (Participants) | 18 | 22
  Week 8 | -18.2 (4.40) | -23.1 (3.59)
Statistical Analysis 1: Comparison: Double-Blind Acute (DBA) Phase: Low Dose vs Double-Blind Acute (DBA) Phase: High Dose; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.168, ANCOVA — P-value is based on an analysis of covariance (ANCOVA) including treatment arm as a factor and baseline DUCS score as a covariate; Difference in Least squares Mean = -5.4, 95% CI 2-sided [-13.1 to 2.4]

6. Secondary Outcome: Number of Participants With Improvement in Pediatric Ulcerative Colitis Activity Index (PUCAI) Score During Double-blind Acute Phase at Week 8
Description: PUCAI was a physician-administered measure that focuses on 6 key signs and symptoms of UC and activity limitations producing a total score ranging from 0-85 with higher scores being worse. Recommended cut-off scores to differentiate disease activity are < 10 (remission); 11-30 (mild); 31-64 (moderate) and > 65 (severe). Participants with an improvement (change of greater than or equal to [> or =] 20 points) in PUCAI score. Number of participants with improvement in PUCAI score during Double-blind Acute Phase at Week 8 were reported.
Time Frame: Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Acute (DBA) Phase: Low Dose | Double-Blind Acute (DBA) Phase: High Dose
Number analyzed (Participants) | 27 | 26
Participants | 10 | 16
Statistical Analysis 1: Comparison: Double-Blind Acute (DBA) Phase: Low Dose vs Double-Blind Acute (DBA) Phase: High Dose; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.131, Chi-squared, Corrected — P-value was based on a continuity-corrected chi-squared test. PUCAI Score was compared between treatment arms using a continuity corrected chi-squared test. Expected cell counts are very low (< 5), then Fisher's Exact Test is alternative method; Difference in proportions = 24.5, 95% CI 2-sided [-1.6 to 50.6]

7. Secondary Outcome: Number of Participants With Clinical and Endoscopic Response During Double-Blind Maintenance Phase at Week 26 Using Central Reading
Description: Clinical and endoscopic response was defined as UC-DAI < or =2 with rectal bleeding=0, stool frequency < or =1, PGA=0, and with mucosal healing (endoscopy score < or =1) based on central reading at Week 26. Number of participants with clinical and endoscopic response during double-blind maintenance phase at Week 26 using central reading were reported.
Time Frame: Week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Maintenance (DBM) Phase: Low Dose | Double-Blind Maintenance (DBM) Phase: High Dose
Number analyzed (Participants) | 42 | 45
Participants | 13 | 11
Statistical Analysis 1: Comparison: Double-Blind Maintenance (DBM) Phase: Low Dose vs Double-Blind Maintenance (DBM) Phase: High Dose; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.539, Cochran-Mantel-Haenszel — P-value is based on a CMH test adjusted by prior response status; Difference in Proportions Percentage = -6.5, 95% CI 2-sided [-25.3 to 12.3]

8. Secondary Outcome: Number of Participants With Clinical and Endoscopic Response During Double-Blind Maintenance Phase at Week 26 Using Local Reading
Description: Clinical and endoscopic response was defined as UC-DAI < or = 2 with rectal bleeding=0, stool frequency < or = 1, PGA=0, and with mucosal healing (endoscopy score < or = 1) based on local reading. Number of participants who had maintained clinical and endoscopic response during double-blind maintenance phase at week 26 using local reading were reported.
Time Frame: Week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Double-Blind Maintenance (DBM) Phase: High Dose: Participants with partial UC-DAI < or =1 and mucosal appearance = 0 or 1 entered the DBM phase directly. Also, participants with a clinical response (partial UC-DAI < or =1) after completion of DBA phase or OLA phase entered into the DBM phase. During the DBM high dose phase participants weighing 18 to < or =23 kg, > 23 to < or =35 kg, > 35 to < or =50 kg, > 50 to < or =90 kg received 1800, 2400, 3600, and 4800 mg/day of MMX mesalamine/mesalazine tablet orally once daily for 26 weeks respectively.
Arm/Group | Double-Blind Maintenance (DBM) Phase: Low Dose | Double-Blind Maintenance (DBM) Phase: High Dose
Number analyzed (Participants) | 42 | 45
Participants | 18 | 12
Statistical Analysis 1: Comparison: Double-Blind Maintenance (DBM) Phase: Low Dose vs Double-Blind Maintenance (DBM) Phase: High Dose; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.129, Cochran-Mantel-Haenszel — P-value was based on a Cochran-Mantel-Haenszel (CMH) test adjusted by prior response status; Difference in proportions = -16.2, 95% CI 2-sided [-36.0 to 3.6]

9. Secondary Outcome: Change From Baseline in Daily Ulcerative Colitis Scale (DUCS) Score During Double-Blind Maintenance Phase
Description: DUCS score was to measure 7 specific signs or symptom and one impact (abdominal pain, nocturnal stool, daytime stool, blood in stool, diarrhea, urgency, tiredness) of UC with each score range from 0 (worst) to 10 (best) with the overall score ranging from 0 (worst) to 70 (best) based on the responses. Change from Baseline in DUCS score during double-blind maintenance phase at week 13 and Week 26 wwere reported.
Time Frame: Baseline, Week 13, and Week 26
Population: Double-blind maintenance phase safety analysis set consisted of randomized participants who had taken at least 1 dose of investigational product during the double-blind maintenance phase. Here, number of participants analyzed signifies participants who were evaluable for this measure category.
Measure: Mean (Standard Error); unit: Score on the scale
Groups:
- Double-Blind Maintenance (DBM) Phase: Low Dose: Participants with partial UC-DAI < or =1 and mucosal appearance = 0 or 1 entered the DBM phase directly. Also, participants with a clinical response (partial UC-DAI < or =1) after completion of DBA phase or OLA phase entered into the DBM phase. During the DBM low dose phase participants weighing 18 to <=23 kg, >23 to <=35 kg, >35 to < or =50 kg, > 50 to < or =90 kg received 900, 1200, 1800, and 2400 mg/day of MMX mesalamine/mesalazine tablet orally once daily for 26 weeks respectively.
Arm/Group | Double-Blind Maintenance (DBM) Phase: Low Dose | Double-Blind Maintenance (DBM) Phase: High Dose
Number analyzed (Participants) | 42 | 45
Score on the scale
  Baseline: number analyzed (Participants) | 41 | 45
  Baseline | 5.8 (1.37) | 4.6 (0.79)
  Week 13: number analyzed (Participants) | 30 | 34
  Week 13 | 1.7 (1.61) | -0.1 (0.89)
  Week 26: number analyzed (Participants) | 26 | 32
  Week 26 | 1.3 (1.19) | 4.4 (1.79)
Statistical Analysis 1: Comparison: Double-Blind Maintenance (DBM) Phase: Low Dose vs Double-Blind Maintenance (DBM) Phase: High Dose; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.182, ANCOVA — P-value was based on an analysis of covariance (ANCOVA) including treatment arm and with prior response status; Difference in Least squares Mean = 3.0, 95% CI 2-sided [-1.4 to 7.4]

10. Secondary Outcome: Number of Participants With Remission at Pediatric Ulcerative Colitis Activity Index (PUCAI) Score During Double-Blind Maintenance Phase at Week 26
Description: PUCAI was a physician-administered measure that focuses on 6 key signs and symptoms of UC and activity limitations producing a total score ranging from 0-85 with higher scores being worse. Recommended cut-off scores to differentiate disease activity are < 10 (remission); 11-30 (mild); 31-64 (moderate) and > 65 (severe). Number of participants with remission at PUCAI score during double-blind maintenance phase at week 26 were reported.
Time Frame: Week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Double-Blind Maintenance (DBM) Phase: High Dose: Participants with partial UC-DAI < or =1 and mucosal appearance = 0 or 1 entered the DBM phase directly. Also, participants with a clinical response (partial UC-DAI < or =1) after completion of DBA phase or OLA phase entered into the DBM phase. During the DBM high dose phase participants weighing 18 to <=23 kg, >23 to <=35 kg, >35 to < or =50 kg, > 50 to < or =90 kg received 1800, 2400, 3600, and 4800 mg/day of MMX mesalamine/mesalazine tablet orally once daily for 26 weeks respectively.
Arm/Group | Double-Blind Maintenance (DBM) Phase: Low Dose | Double-Blind Maintenance (DBM) Phase: High Dose
Number analyzed (Participants) | 42 | 45
Participants | 29 | 27
Statistical Analysis 1: Comparison: Double-Blind Maintenance (DBM) Phase: Low Dose vs Double-Blind Maintenance (DBM) Phase: High Dose; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.194, Cochran-Mantel-Haenszel — P-value was based on a CMH test adjusted by prior response status. Participants with remission (PUCAI <10) at double-blind maintenance phase at Week 26 was compared between treatment arms using a CMH test stratifying by Week 8 responder status; Difference in proportions = -9.0, 95% CI 2-sided [-29.1 to 11.0]

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (up to Week 27)
Description: Overall safety analysis set consisted of randomized participants who had taken at least 1 dose of IP.
Groups:
- Double-Blind Acute (DBA) Phase: Low Dose: Participants with partial UC-DAI >=2 and mucosal appearance = 2 or 3 entered the DBA phase. During the DBA low dose phase participants weighing 18 to <=23 kg, >23 to <=35 kg, >35 to <=50 kg, >50 to <=90 kg received 900, 1200, 1800, and 2400 mg/day of MMX mesalamine/mesalazine tablet orally once daily for 8 weeks respectively.
- Double-Blind Acute (DBA) Phase: High Dose: Participants with partial UC-DAI >=2 and mucosal appearance = 2 or 3 entered the DBA phase. During the DBA high dose phase participants weighing 18 to <=23 kg, >23 to <=35 kg, >35 to <=50 kg, >50 to <=90 kg received 1800, 2400, 3600, and 4800 mg/day of MMX mesalamine/mesalazine tablet orally once daily for 8 weeks respectively.
- Open-Label Acute (OLA) Phase: High Dose: Participants with partial UC-DAI between 1 and 2 entered the OLA phase, after completing DBA phase. Participants weighing 18 to <=23 kg, >23 to <=35 kg, >35 to <=50 kg, >50 to <=90 kg received 1800, 2400, 3600, and 4800 mg/day of MMX mesalamine/mesalazine tablet orally once daily for 8 weeks respectively during the high dose OLA phase.
- Double-Blind Maintenance (DBM) Phase: Low Dose: Participants with partial UC-DAI <=1 and mucosal appearance = 0 or 1 entered the DBM phase directly. Also, participants with a clinical response (partial UC-DAI <=1) after completion of DBA phase or OLA phase entered into the DBM phase. During the DBM low dose phase participants weighing 18 to <=23 kg, >23 to <=35 kg, >35 to <=50 kg, >50 to <=90 kg received 900, 1200, 1800, and 2400 mg/day of MMX mesalamine/mesalazine tablet orally once daily for 26 weeks respectively.
- Double-Blind Maintenance (DBM) Phase: High Dose: Participants with partial UC-DAI <=1 and mucosal appearance = 0 or 1 entered the DBM phase directly. Also, participants with a clinical response (partial UC-DAI <=1) after completion of DBA phase or OLA phase entered into the DBM phase. During the DBM high dose phase participants weighing 18 to <=3 kg, >23 to <=35 kg, >35 to <=50 kg, >50 to <=90 kg received 1800, 2400, 3600, and 4800 mg/day of MMX mesalamine/mesalazine tablet orally once daily for 26 weeks respectively.
Arm/Group | Double-Blind Acute (DBA) Phase: Low Dose | Double-Blind Acute (DBA) Phase: High Dose | Open-Label Acute (OLA) Phase: High Dose | Double-Blind Maintenance (DBM) Phase: Low Dose | Double-Blind Maintenance (DBM) Phase: High Dose
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26 | 0/18 | 0/42 | 0/45
Serious Adverse Events (participants affected / at risk) | 4/27 | 0/26 | 3/18 | 3/42 | 2/45
Other Adverse Events (participants affected / at risk) | 15/27 | 15/26 | 12/18 | 25/42 | 25/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Acute (DBA) Phase: Low Dose (N=27) | Double-Blind Acute (DBA) Phase: High Dose (N=26) | Open-Label Acute (OLA) Phase: High Dose (N=18) | Double-Blind Maintenance (DBM) Phase: Low Dose (N=42) | Double-Blind Maintenance (DBM) Phase: High Dose (N=45)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Colitis ulcerative (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury corneal (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Acute (DBA) Phase: Low Dose (N=27) | Double-Blind Acute (DBA) Phase: High Dose (N=26) | Open-Label Acute (OLA) Phase: High Dose (N=18) | Double-Blind Maintenance (DBM) Phase: Low Dose (N=42) | Double-Blind Maintenance (DBM) Phase: High Dose (N=45)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (5) | 5 (6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 6 (6) | 0 (0) | 1 (1) | 5 (5) | 8 (9)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (8)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 6 (6)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (3) | 2 (6)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT02093663/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT02093663/SAP_001.pdf